CLINICAL TRIAL: NCT05168410
Title: Sensitivity and Specificity of the Alvarado Score for the Timely Differential Diagnosis of Acute Appendicitis in Samoa
Status: Completed | Type: Observational
Sponsor: Dr Annette Kaspar (Other Government)
Collaborators: Fiji National University (Other)
Responsible Party: Sponsor-Investigator, Dr Annette Kaspar, Head of Audiology, Tupua Tamasese Meaole Hospital
Organization: Tupua Tamasese Meaole Hospital (Other Government)
Other Study IDs: s994956
Record Dates: First submitted 2021-11-14; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Acute Appendicitis
Keywords: Alvarado Score
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Alvarado Score — The Alvarado Score assesses patient symptoms to enable optimal triage and management of cases with suspected acute appendicitis.a

SUMMARY:
Retrospective clinical data review design of all patients admitted to the Tupua Tamasese Meaole Hospital Surgical Unit for AA from January 2015 to December 2016. Exclusion criteria were appendiceal abscess and/or mass, and final diagnosis 'not acute appendicitis'. Age, sex, village, Alvarado Score, Ultrasound Scan Result, surgical management, and histopathology result were the main variables entered into the SPSS statistical software package for analysis.

DETAILED DESCRIPTION:
METHODS

Study Design and Data Collection

A retrospective study design was used to evaluate all AA cases seen by the Surgical Department of TTM Hospital over the 24-month period between 1 January 2015 and 31 December 2016. The clinical medical records were obtained from the National Health Service PATIS System, using the search terms 'appendicitis', 'acute appendicitis', and 'appendicectomy'. A total of 289 records were retrieved. Thirty four (34) records were excluded having met the exclusion criteria: (1) final diagnosis was not AA (i.e., ectopic pregnancy, tubal ovarian abscess, other gynaecological pathologies, diverticulitis, Merkel diverticulitis, perforated ulcer), and (2) appendiceal abscess and/or appendiceal mass. Thirty (30) clinical records with missing data, and these were also excluded from the study. The final number of included for analysis was 225 cases. All 225 cases were initially treated with intravenous antibiotics upon presentation to the emergency department as per the National Health Service antibiotic guidelines: intravenous ceftriaxone and metronidazole was the first line of treatment, and alternative antibiotics were administered if unavailable (i.e., clindamycin + gentamycin or ampicillin, or gentamycin + metronidazole).

A purpose-designed data collection form and excel spreadsheet were created for the study. The following information was extracted from the clinical records: patient gender (male/female), age (years), address (urban/rural), time of admission (Morning/Afternoon/Night Shift), use of traditional/alternative medicine prior to attending emergency department (yes/no), administration of antibiotics by emergency department staff (yes/no), Alvarado Score (1-10), Ultrasound Scan for AA (Positive/negative/Inconclusive/Not performed), management of AA (appendicectomy/antibiotic therapy), intra-operative macroscopic examination (Grade 1-5), histopathology result for AA (Positive/Negative/Inconclusive/Not available), length of stay in hospital (days), and mortality (yes/no).

Data analysis The data was analysed using the SPSS (Version 2.1) statistical software package. Descriptive analysis was performed, and the chi-square test of significance was used to investigate for statistically significant differences between variables (significant at p<0.05). The sensitivity, specificity, Positive Predictive Value (PPV), and Negative Predictive Value (NPV) were calculated for the Alvarado Score in identifying AA as confirmed by histopathology.

ELIGIBILITY:
Inclusion Criteria:

• All Acute Appendicitis (AA) cases seen by the Surgical Department of TTM Hospital over the 24-month period between 1 January 2015 and 31 December 2016.

Exclusion Criteria:

* Final diagnosis was not Acute Appendicitis (i.e., ectopic pregnancy, tubal ovarian abscess, other gynaecological pathologies, diverticulitis, Merkel diverticulitis, perforated ulcer)
* Final diagnosis was appendiceal abscess and/or appendiceal mass.
* Clinical records with missing data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Acute Appendicitis cases seen by the Surgical Department of TTM Hospital over the 24-month period between 1 January 2015 and 31 December 2016.
  The final number of included for analysis was 225 cases.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the Alvarado Score for the identification of acute appendicitis in Samoa | 24 months
  The sensitivity of the Alvarado Score will be calculated for correct diagnosis of acute appendicitis based on confirmed acute appendicitis by histopathology results

SECONDARY OUTCOMES:
Accuracy of the Alvarado Score for the identification of acute appendicitis in Samoa | 24 months
  The specificity of the Alvarado Score will be calculated for correct diagnosis of acute appendicitis based on confirmed cases of acute appendicitis by histopathology

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.